CLINICAL TRIAL: NCT02749110
Title: Participation in Screening for Cervical Cancer: Interest of a Human Papillomavirus (HPV) Self-sampling Device Provided by the General Practitioner; a Cluster Randomized Clinical Trial
Brief Title: Participation in Screening for Cervical Cancer: Interest of a Self-sampling Device Provided by the General Practitioner
Acronym: PaCUDAHL-Gé
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015_08; 2015-A01331-48 (Other: ID-RCB number, ANSM); LIC-14-14-0615 (Other: PREPS number, DGOS)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2020-08

CONDITIONS: Malignant Tumor of Cervix; Cervical Intraepithelial Neoplasia
Keywords: Mass screening; Family medicine; Human Papillomavirus DNA tests; Papanicolaou test; Early detection of cancer/methods*; Specimen Handling/methods*; Patient compliance; Adult; Female; Humans; Randomized controlled trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-sampling for HPV test (Experimental): Invitation to participate to the screening process by means of the usual care (pap-test) or the provision of a vaginal self-sampling brush (Evalyn Brush°). Self-collected samples are mailed to a central lab for HPV testing.
  Interventions: Device: Vaginal self-sampling brush
- Usual care (Pap test) (No Intervention): Intervention: invitation to participate to the screening process by means of the usual care (pap-test).

INTERVENTIONS:
Device: Vaginal self-sampling brush — Self-collection by unscreened women aged from 30 to 65 of a vaginal sample with the device. After collection, the whole device is mailed in a normalized for biological samples package to the virology lab of the University Hospital of Lille where a HPV test is conducted using a Cobas 4800 technique.
  Other Names: Evalyn Brush; European Community (EC) certificate N°: 44232121392
  Arms: Self-sampling for HPV test

SUMMARY:
This study evaluates the benefit in women aged from 30 to 65 years, who do not participate to the French opportunistic cervical cancer screening program, of an organized screening with the proposition by the family physician of a pap-test (usual care) versus a self-collected vaginal sample (and a HPV-test). 24 family physicians will participate and will be randomized in the usual care arm (12) or in the self-sampling arm (12). Our hypothesis is that organizing the screening for these women involving their family physician will major participation, and that the self-sampling option will amplify this increase.

DETAILED DESCRIPTION:
In France screening for cervical cancer (CC) is usually based on an opportunistic screening program. French guidance recommends performing a smear every 3 years from the age of 25 to 65 years, after 2 initial normal yearly smears. Pap-tests can be carried out by medical doctors or midwifes. The coverage rate is estimated between 56.6% and 83.0%. In deprived populations, about 55% of women are unscreened as their risk to develop a CC is majored. The gynecologic examination and the consultation of a gynecologist appear to be the main barriers to the pap-test. Almost all these unscreened women visit their family physician at least yearly for themselves or with a relative, but many family physicians do not perform pap-tests. Our hypothesis is that more women are to be screened if they are invited to by their family physician (who carries out the pap-test himself or who refers the woman to a gynecologist or a midwife), and that the screening rate will be majored if the family physician delivers to his female patients, who are not willing to undergo a pap-smear, a vaginal self-sampling device.

To demonstrate this, we will conduct an open label 1:1 cluster randomized controlled trial. As the gender of the physician and his ability to carry out pap-tests is associated to the rate of his listed screened female patients, randomization will be stratified on these two variables. The 24 participating physicians (12 in each study arm) will enroll 2000 unscreened female patients. The study population will be all the social security insured unscreened listed women aged from 30 to 65 years of the participating physicians. As the specificity of the HPV-test to screen for CC is insufficient before the age of 30, woman between 25 and 29 years of age will not be part of the study.

All these women (unless an exclusion criterion appears in their medical record) will receive from their family physician an invitation letter to make an appointment for an encounter dedicated to CC screening. Women who accept to be enrolled in the study will sign a consent form and will be invited to fill in a questionnaire about their socio-economic profile and their beliefs and attitudes about prevention, cancer screening in general and screening for CC in particular. Participation to the screening process is not necessary for inclusion. Women in the control arm will be solely proposed to undergo a pap-test performed by their family physician or a gynecologist or a midwife. Women in the intervention arm will be alternatively proposed to proceed to an at home performed vaginal self-collection of a sample that is to be send by post to a centralized lab for HPV testing. HPV tests will be conducted by the virology lab of the University Hospital of Lille.

All screened negative women in both arms of the study will be considered as successful outcomes and finish the study. HPV screened positive women from the self-collection arm will be proposed a triage pap-test or colposcopy. Further 18 months follow-up will be matching French guidelines.

ELIGIBILITY:
Inclusion Criteria:

* To be a woman
* Aged from 30 to 65 years (30 and 65 years included)
* Without reimbursement of a pap-test by the health insurance for more than 3 years, despite a reminder mailed by the health insurance on the previous year (list set up by the health insurance).
* Able to understand and sign voluntarily the consent to participate
* Warranted by the health insurance
* Able to understand and answer the questions of the study questionnaire alone or with the help of a self-chosen third party.

Exclusion Criteria:

* No vaginal intercourse ever
* Pap-test quoted on another budget (hospital, mother and child protection…) conducted less than 3 years ago
* Known cervical lesion or known HPV status
* History of hysterectomy
* History of conisation
* History of laser treatment of the cervix
* History of cervical cancer
* Other medical reason to delay cervical cancer screening
* Abroad for more than one year
* Moving to another region (done or expected)
* Pregnant or breastfeeding
* Screening not relevant from the practitioner's perspective (Emergency situation, comorbidity…)

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2016-08-28 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Rate of women terminating the whole diagnostic process. | For screening: 12 months; for follow-up of screened positive subjets: 18 months
  Women participating in the study but refusing the screening process are considered as "failure

SECONDARY OUTCOMES:
Theory of planned behavior (TPB) see Ajzen-Fishbein | At baseline
  Data collected by self-completed questionnaire.psychological determinants of screening in 7 groups of variables (Attitudes, norms, Self-efficacy, intention, environmental factors, skills and abilities, behavior)
social determinants of screening (age, level of education, level of resources, vocational situation, matrimonial status…) | At baseline
  Data collected by self-completed questionnaire

OTHER OUTCOMES:
European Deprivation Index (EDI) associated to the dwelling of the study subjects | At baseline
  The EDI is an index based on 8 demographic determinants

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Berkhout, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Doctor's office 115, Herzeele, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fishbein M. A reasoned action approach to health promotion. Med Decis Making. 2008 Nov-Dec;28(6):834-44. doi: 10.1177/0272989X08326092. Epub 2008 Nov 17. PMID 19015289
- [Background] van Baars R, Bosgraaf RP, ter Harmsel BW, Melchers WJ, Quint WG, Bekkers RL. Dry storage and transport of a cervicovaginal self-sample by use of the Evalyn Brush, providing reliable human papillomavirus detection combined with comfort for women. J Clin Microbiol. 2012 Dec;50(12):3937-43. doi: 10.1128/JCM.01506-12. Epub 2012 Sep 26. PMID 23015677
- [Background] Viguier J, Calazel-Benque A, Eisinger F, Pivot X. Organized colorectal cancer screening programmes: how to optimize efficiency among general practitioners. Eur J Cancer Prev. 2011 Jan;20 Suppl 1:S26-32. doi: 10.1097/01.cej.0000391567.49006.af. PMID 21245677
- [Background] Verhoef VM, Bosgraaf RP, van Kemenade FJ, Rozendaal L, Heideman DA, Hesselink AT, Bekkers RL, Steenbergen RD, Massuger LF, Melchers WJ, Bulten J, Overbeek LI, Berkhof J, Snijders PJ, Meijer CJ. Triage by methylation-marker testing versus cytology in women who test HPV-positive on self-collected cervicovaginal specimens (PROHTECT-3): a randomised controlled non-inferiority trial. Lancet Oncol. 2014 Mar;15(3):315-22. doi: 10.1016/S1470-2045(14)70019-1. Epub 2014 Feb 13. PMID 24529697
- [Background] Duport N, Serra D, Goulard H, Bloch J. [Which factors influence screening practices for female cancer in France?]. Rev Epidemiol Sante Publique. 2008 Oct;56(5):303-13. doi: 10.1016/j.respe.2008.07.086. Epub 2008 Oct 31. French. PMID 18951740
- [Result] Favre J, Rochoy M, Raginel T, Pelletier M, Messaadi N, Deken-Delannoy V, Duhamel A, Berkhout C. The Effect of Cervical Smears Performed by General Practitioners on the Cervical Cancer Screening Rate of their Female Patients: A Claim Database Analysis and Cross-Sectional Survey. J Womens Health (Larchmt). 2018 Jul;27(7):933-938. doi: 10.1089/jwh.2017.6656. Epub 2018 Mar 27. PMID 29583084
- [Result] Anhang R, Nelson JA, Telerant R, Chiasson MA, Wright TC Jr. Acceptability of self-collection of specimens for HPV DNA testing in an urban population. J Womens Health (Larchmt). 2005 Oct;14(8):721-8. doi: 10.1089/jwh.2005.14.721. PMID 16232104
- [Result] Haguenoer K, Giraudeau B, Gaudy-Graffin C, de Pinieux I, Dubois F, Trignol-Viguier N, Viguier J, Marret H, Goudeau A. Accuracy of dry vaginal self-sampling for detecting high-risk human papillomavirus infection in cervical cancer screening: a cross-sectional study. Gynecol Oncol. 2014 Aug;134(2):302-8. doi: 10.1016/j.ygyno.2014.05.026. Epub 2014 Jun 3. PMID 24905772
- [Result] Cadman L, Ashdown-Barr L, Waller J, Szarewski A. Attitudes towards cytology and human papillomavirus self-sample collection for cervical screening among Hindu women in London, UK: a mixed methods study. J Fam Plann Reprod Health Care. 2015 Jan;41(1):38-47. doi: 10.1136/jfprhc-2013-100705. Epub 2014 Feb 12. PMID 24521934
- [Result] Waller J, Bartoszek M, Marlow L, Wardle J. Barriers to cervical cancer screening attendance in England: a population-based survey. J Med Screen. 2009;16(4):199-204. doi: 10.1258/jms.2009.009073. PMID 20054095
- [Result] Cox JT, Castle PE, Behrens CM, Sharma A, Wright TC Jr, Cuzick J; Athena HPV Study Group. Comparison of cervical cancer screening strategies incorporating different combinations of cytology, HPV testing, and genotyping for HPV 16/18: results from the ATHENA HPV study. Am J Obstet Gynecol. 2013 Mar;208(3):184.e1-184.e11. doi: 10.1016/j.ajog.2012.11.020. Epub 2012 Nov 19. PMID 23174289
- [Result] Park Y, Lee E, Choi J, Jeong S, Kim HS. Comparison of the Abbott RealTime High-Risk Human Papillomavirus (HPV), Roche Cobas HPV, and Hybrid Capture 2 assays to direct sequencing and genotyping of HPV DNA. J Clin Microbiol. 2012 Jul;50(7):2359-65. doi: 10.1128/JCM.00337-12. Epub 2012 Apr 18. PMID 22518863
- [Result] TOMBOLA Group. Cytological surveillance compared with immediate referral for colposcopy in management of women with low grade cervical abnormalities: multicentre randomised controlled trial. BMJ. 2009 Jul 28;339:b2546. doi: 10.1136/bmj.b2546. PMID 19638646
- [Result] Rigal L, Saurel-Cubizolles MJ, Falcoff H, Bouyer J, Ringa V. Do social inequalities in cervical cancer screening persist among patients who use primary care? The Paris Prevention in General Practice survey. Prev Med. 2011 Sep;53(3):199-202. doi: 10.1016/j.ypmed.2011.06.016. Epub 2011 Jun 25. PMID 21726576
- [Result] Chan Chee C, Begassat M, Kovess V. [Factors associated with cervical cancer screening in women covered by national health insurance]. Rev Epidemiol Sante Publique. 2005 Feb;53(1):69-75. doi: 10.1016/s0398-7620(05)84573-0. French. PMID 15888991
- [Result] Zehbe I, Moeller H, Severini A, Weaver B, Escott N, Bell C, Crawford S, Bannon D, Paavola N. Feasibility of self-sampling and human papillomavirus testing for cervical cancer screening in First Nation women from Northwest Ontario, Canada: a pilot study. BMJ Open. 2011 Feb 26;1(1):e000030. doi: 10.1136/bmjopen-2010-000030. PMID 22021733
- [Result] Goodman A. HPV testing as a screen for cervical cancer. BMJ. 2015 Jun 30;350:h2372. doi: 10.1136/bmj.h2372. PMID 26126623
- [Result] Gok M, Heideman DA, van Kemenade FJ, Berkhof J, Rozendaal L, Spruyt JW, Voorhorst F, Belien JA, Babovic M, Snijders PJ, Meijer CJ. HPV testing on self collected cervicovaginal lavage specimens as screening method for women who do not attend cervical screening: cohort study. BMJ. 2010 Mar 11;340:c1040. doi: 10.1136/bmj.c1040. PMID 20223872
- [Result] Broberg G, Gyrd-Hansen D, Miao Jonasson J, Ryd ML, Holtenman M, Milsom I, Strander B. Increasing participation in cervical cancer screening: offering a HPV self-test to long-term non-attendees as part of RACOMIP, a Swedish randomized controlled trial. Int J Cancer. 2014 May 1;134(9):2223-30. doi: 10.1002/ijc.28545. Epub 2013 Oct 31. PMID 24127304
- [Result] Grillo F, Vallee J, Chauvin P. Inequalities in cervical cancer screening for women with or without a regular consulting in primary care for gynaecological health, in Paris, France. Prev Med. 2012 Mar-Apr;54(3-4):259-65. doi: 10.1016/j.ypmed.2012.01.013. Epub 2012 Jan 24. PMID 22296836
- [Result] Elfstrom KM, Smelov V, Johansson AL, Eklund C, Naucler P, Arnheim-Dahlstrom L, Dillner J. Long term duration of protective effect for HPV negative women: follow-up of primary HPV screening randomised controlled trial. BMJ. 2014 Jan 16;348:g130. doi: 10.1136/bmj.g130. PMID 24435414
- [Result] Gok M, Heideman DA, van Kemenade FJ, de Vries AL, Berkhof J, Rozendaal L, Belien JA, Overbeek L, Babovic M, Snijders PJ, Meijer CJ. Offering self-sampling for human papillomavirus testing to non-attendees of the cervical screening programme: Characteristics of the responders. Eur J Cancer. 2012 Aug;48(12):1799-808. doi: 10.1016/j.ejca.2011.11.022. Epub 2011 Dec 13. PMID 22172570
- [Result] Bulk S, Bulkmans NW, Berkhof J, Rozendaal L, Boeke AJ, Verheijen RH, Snijders PJ, Meijer CJ. Risk of high-grade cervical intra-epithelial neoplasia based on cytology and high-risk HPV testing at baseline and at 6-months. Int J Cancer. 2007 Jul 15;121(2):361-7. doi: 10.1002/ijc.22677. PMID 17354241
- [Result] Lazcano-Ponce E, Lorincz AT, Cruz-Valdez A, Salmeron J, Uribe P, Velasco-Mondragon E, Nevarez PH, Acosta RD, Hernandez-Avila M. Self-collection of vaginal specimens for human papillomavirus testing in cervical cancer prevention (MARCH): a community-based randomised controlled trial. Lancet. 2011 Nov 26;378(9806):1868-73. doi: 10.1016/S0140-6736(11)61522-5. Epub 2011 Nov 1. PMID 22051739
- [Result] Cullen J, Schwartz MD, Lawrence WF, Selby JV, Mandelblatt JS. Short-term impact of cancer prevention and screening activities on quality of life. J Clin Oncol. 2004 Mar 1;22(5):943-52. doi: 10.1200/JCO.2004.05.191. PMID 14990651
- [Result] C Kitchener H, Canfell K, Gilham C, Sargent A, Roberts C, Desai M, Peto J. The clinical effectiveness and cost-effectiveness of primary human papillomavirus cervical screening in England: extended follow-up of the ARTISTIC randomised trial cohort through three screening rounds. Health Technol Assess. 2014 Apr;18(23):1-196. doi: 10.3310/hta18230. PMID 24762804
- [Result] Giorgi Rossi P, Marsili LM, Camilloni L, Iossa A, Lattanzi A, Sani C, Di Pierro C, Grazzini G, Angeloni C, Capparucci P, Pellegrini A, Schiboni ML, Sperati A, Confortini M, Bellanova C, D'Addetta A, Mania E, Visioli CB, Sereno E, Carozzi F; Self-Sampling Study Working Group. The effect of self-sampled HPV testing on participation to cervical cancer screening in Italy: a randomised controlled trial (ISRCTN96071600). Br J Cancer. 2011 Jan 18;104(2):248-54. doi: 10.1038/sj.bjc.6606040. Epub 2010 Dec 21. PMID 21179038
- [Derived] Rochoy M, Raginel T, Favre J, Soueres E, Messaadi N, Deken V, Duhamel A, Berkhout C. Factors associated with the achievement of cervical smears by general practitioners. BMC Res Notes. 2017 Dec 8;10(1):723. doi: 10.1186/s13104-017-2999-5. PMID 29221494